CLINICAL TRIAL: NCT00386750
Title: An Open-label, Single-center Study of the Effects of Co-artemether, Atovaquone-proguanil, and Artesunate-mefloquine on Auditory Function Following the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Patients 12 Years of Age or Older.
Brief Title: Safety of Artemether - Lumefantrine, and Other Malaria Drugs and Their Effect on the Auditory Function
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566A2412
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Malaria; Falciparum
Keywords: Malaria; hearing; co-artemether; auditory; Plasmodium falciparum; marsh fever; Plasmodium infections; remittent fever; paludism; artemether; artemisinins; benflumetol; lumefantrine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Artemether-lumefantrine

SUMMARY:
THIS STUDY IS NOT ENROLLING PATIENTS IN THE USA.

To evaluate the effects of artemether/ lumefantrine on the auditory function.

ELIGIBILITY:
Inclusion Criteria

* 12 years of age or older
* P. falciparum parasitemia between 50 and 100,000 parasites/μl
* History of fever or presence of fever (temperature ≥ 37.5°C)

Exclusion Criteria

* Signs/symptoms of severe/complicated malaria
* Ingestion of various antimalarial drugs, or antibiotics in the previous 2 weeks to 2 months
* History of any drug-related hearing impairment.
* Abnormal hearing function at study entry
* Exposure to sustained loud noises, by self-report, within the past 24 hours. -- Present ear problems

(Other protocol-defined inclusion/exclusion criteria may apply.)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265
Dates: Start 2005-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Auditory abnormalities at Day 7 assessed by Auditory Brainstem Response (ABR) wave form latencies (a type of hearing test).

SECONDARY OUTCOMES:
Rate of auditory changes following 3 days of treatment with artemether-lumefantrine at Days 7, 28, and 42 days assessed by pure tone thresholds assessments (a type of hearing test)
Changes in auditory function with a non-ACT (artemisinin combined therapy) antimalarial (Malarone, atovaquone-proguanil) and another ACT combination (artesunate-mefloquine) assessed by pure tone thresholds (a type of hearing test)
Relationship between changes in auditory function and drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals